CLINICAL TRIAL: NCT06351735
Title: Evaluation of the Efficacy and Safety of Deep Cervical Lymph Node-vein Bypass Surgery in Patients With Amyotrophic Lateral Sclerosis
Brief Title: Efficacy and Safety of Deep Cervical Lymph Node-vein Bypass Surgery in ALS Amyotrophic Lateral Sclerosis
Status: Not yet recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Yuanjian Fang, Principal Investigator, Second Affiliated Hospital, School of Medicine, Zhejiang University
Other Study IDs: 2024-0336
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Efficacy and Safety
Keywords: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cerebrospinal fluid and blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgery: Patients undergo deep cervical lymph node-vein bypass surgery
  Interventions: Procedure: Deep cervical lymph node-vein bypass surgery

INTERVENTIONS:
Procedure: Deep cervical lymph node-vein bypass surgery — Deep cervical lymph node-vein bypass surgery, connecting deep cervical lymph node input lymphatic vessel

SUMMARY:
Amyotrophic lateral sclerosis (ALS), a fatal neurodegenerative disease, affects motor neurons, causing progressive muscle atrophy and weakness. Current treatments are ineffective, with most patients dying within 3-5 years of diagnosis. The disease's exact cause is unclear, but factors such as oxidative stress and protein abnormalities are implicated. Abnormal protein deposits and neurotoxic factors in the brain and spinal cord contribute to ALS pathology. Recent research on the brain's glymphatic-lymphatic system suggests impaired waste clearance may exacerbate ALS. Restoring drainage connections between cervical lymphatic vessels and veins could potentially alleviate neurodegenerative disease progression.

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis (ALS) is a fatal neurodegenerative disease characterized by the simultaneous involvement of upper and lower motor neurons, leading to progressive muscle atrophy and weakness in patients. Advanced stages of the disease manifest as symptoms such as swallowing difficulties and respiratory problems. Currently, effective treatments for ALS are lacking, and most patients succumb to the disease within 3 to 5 years of onset. Therefore, there is an urgent need to explore new therapeutic approaches. Although the exact pathogenesis of ALS remains unclear, various mechanisms including oxidative stress, glutamate toxicity, mitochondrial dysfunction, endoplasmic reticulum stress, and protein misfolding are thought to contribute to its development. Pathological findings indicate the presence of abnormal protein deposits, including phosphorylated TDP-43 (Transactive response DNA-binding protein 43 kDa), superoxide dismutase 1 (SOD1), and dysfunctional ribosomal proteins, in the brains and spinal cords of ALS patients. Additionally, elevated levels of neurotoxic factors in the cerebrospinal fluid, such as inflammatory cytokines and reactive oxygen species, have been implicated in the pathogenesis of ALS. Therefore, clearance of abnormal proteins and neurotoxic factors from the brain and spinal cord may have potential therapeutic implications for delaying or preventing neurodegeneration and associated clinical disabilities in ALS patients.

Recently, the discovery of the brain "glymphatic-lymphatic" system has updated our understanding of cerebrospinal fluid circulation. Similar to the peripheral lymphatic circulation, there exists an interstitial fluid circulation system in the brain parenchyma. Studies have revealed that cerebrospinal fluid in the brain parenchyma enters the perivascular spaces surrounding arteries through aquaporin-4 channels on astrocytes and then flows directionally into the perivascular spaces surrounding veins, facilitating waste clearance and nutrient transport in the brain. This phenomenon is known as the glymphatic system. Furthermore, abundant lymphatic vessels have been found adjacent to the dural venous sinuses, participating in cerebrospinal fluid drainage and ultimately draining into the cervical lymph nodes. In animal models of Alzheimer's disease (AD) and Parkinson's disease (PD), impairment of the glymphatic-lymphatic drainage function has been associated with the accumulation of disease-related proteins such as amyloid beta (Aβ), Tau, and alpha-synuclein, and ligating the cervical lymph nodes has been shown to exacerbate disease progression. Clinical studies using magnetic resonance imaging have confirmed the decline in glymphatic-lymphatic system function in patients with AD and PD. Although research on the role and mechanism of the glymphatic-lymphatic drainage system in the occurrence and development of ALS is lacking, magnetic resonance imaging has revealed a significant reduction in glymphatic system function in ALS patients compared to healthy individuals, suggesting an important role of the glymphatic-lymphatic drainage system in the pathogenesis of ALS.

As the final destination of glymphatic-lymphatic cerebrospinal fluid drainage, the cervical lymph nodes play a crucial role in the entire cerebrospinal fluid circulation. With aging, infection, and chronic inflammation, the function of the cervical lymph nodes gradually declines, leading to increased cerebrospinal fluid circulation reflux pressure. Furthermore, the production of large amounts of neurotoxic substances during the progression of AD, PD, and ALS further impairs the function of the cervical lymph nodes, resulting in abnormal accumulation of toxic substances in the brain and disease progression. We speculate that establishing drainage connections between the cervical lymphatic vessels and veins will reduce cerebrospinal fluid circulation pressure in brain tissues, accelerate interstitial fluid reflux, and alleviate the accumulation of metabolic waste, thereby slowing the progression of neurodegenerative diseases.

ELIGIBILITY:
Inclusion Criteria:

* ①diagnosis of probable, clinically probable, clinically probable laboratory-supported, or clinically definite ALS according to the revised El Escorial World Federation of Neurology criteria; ② aged between 20 and 80 years old (inclusive); ③ ALS patients with King's Stage 3-4; ④ body weight not less than 45 kg and body mass index (BMI) not less than 18.0 kg/m2; 5) not currently receiving riluzole or receiving a stable dose of riluzole for at least 4 weeks before screening; Subjects who received riluzole were expected to maintain the same dose throughout the study; ⑦ Subjects' FVC≥60% predicted value after adjusting for sex, age, and height.

Exclusion Criteria:

* ① Refusal to participate; ② Unable to complete MRI scan; ③ significant cognitive impairment, mental illness, epilepsy or other neurodegenerative diseases, substance abuse; ④ recent severe infection or infectious diseases within 4 weeks; ⑤ complicated with other systemic underlying diseases; Any past stem cell or gene therapy for ALS.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ALS patients meet to the inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 3 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
ALSFRS-R scale | Pre-surgery and post-surgery 1month, 3 months, 6 months and 1 year
  Improvement of ALSFRS-R scale
Cognitive and Behavioral Scale (CAS) | Pre-surgery and post-surgery 1month, 3 months, 6 months and 1 year
  Improvement of CAS score

SECONDARY OUTCOMES:
Baseline of slow vital capacity (SVC) | Pre-surgery and post-surgery 1month, 3 months, 6 months and 1 year
  Change baseline of SVC
Evaluation of glymphatic and meningeal lymphatic drainage | Pre-surgery and post-surgery 3 months, 6 months and 1 year
  MRI evaluation of glymphatic and meningeal lymphatic drainage
Amyotrophic Lateral Sclerosis Assessment Questionnaire (ALSAQ-5) | Pre-surgery and post-surgery 3 months, 6 months and 1 year
  Changes from baseline in the Amyotrophic Lateral Sclerosis Assessment Questionnaire (ALSAQ-5)

IPD SHARING:
Plan to Share IPD: No